CLINICAL TRIAL: NCT04742595
Title: Administration of Expanded, Most Closely HLA Matched SARS-CoV-2-Specific T Cells for the Treatment of COVID-19 in Patients With Cancer
Brief Title: Viral Specific T Cell Therapy for COVID-19 Related Pneumonia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0759; NCI-2020-13875 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0759 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SARS-COV-2 specific cytotoxic T cells) (Experimental): Patients receive SARS-COV-2 specific cytotoxic T lymphocytes IV over 30 minutes on day 1. Treatment may repeat every 14 days at investigators' discretion if patient fails to respond, the infection reoccurs, until the viral load becomes negative or until complete resolution of clinical and radiological signs.
  Interventions: Biological: SARS-CoV-2 Antigen-specific Cytotoxic T-lymphocytes

INTERVENTIONS:
Biological: SARS-CoV-2 Antigen-specific Cytotoxic T-lymphocytes — Given IV
  Other Names: SARS-CoV-2 Antigen-specific CTLs; SARS-CoV-2 Antigen-specific Cytotoxic T Lymphocytes; SARS-CoV-2-specific Cytotoxic T-lymphocytes

SUMMARY:
This early phase I trial identifies the feasibility, possible benefits and/or side effects of administering SARS-CoV-2 specific cytotoxic T lymphocytes (CTLs) in treating cancer patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, the virus responsible for coronavirus disease 2019 (COVID-19). SARS-CoV-2 Specific CTLs are a type of immune cells that are made from donated blood cells grown in the laboratory and are designed to kill cells infected with SARS-CoV-2 virus. Giving CTLs may help control the COVID-19 in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and safety of administering most closely human leukocyte antigen (HLA)-matched severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) specific T cell lines generated by ex vivo expansion as therapy of COVID19 pneumonia in cancer patients.

SECONDARY OBJECTIVES:

I. To obtain preliminary data about the efficacy of administering most closely HLA-matched SARS-COV-2 specific T cell lines generated by ex vivo expansion.

II. To assess the persistence of the administered cells in the patients.

OUTLINE:

Patients receive SARS-COV-2 specific cytotoxic T lymphocytes intravenously (IV) over 30 minutes on day 1. Treatment may repeat every 14 days at investigators' discretion if patient fails to respond, the infection reoccurs, until the viral load becomes negative or until complete resolution of clinical and radiological signs.

After completion of study treatment, patients are followed up at 7, 14, 21, 28, and 45 days, and 3 months after each cytotoxic T lymphocyte infusion.

ELIGIBILITY:
Inclusion criteria:

Immunocompromised patients with hematological malignances and diagnosis of COVID-19 > 3 weeks prior to study entry, treated with at least one SOC therapy (i.e., remdesivir, monoclonal antibody [bebtelovimab or newer one], paxlovid, molnupiravir, corticosteroids, other EUA or FDA-approved therapies) with progression of symptoms in the following 14 days after treatment started, of at least 1 category on the 8 ordinal category on the 8 ordinal category WHO scale, or CT chest/CXR shows progression of pneumonia or increase oxygen requirements of at least 2 liters from baseline. Patients should not show signs of improvement before enrollment.

* World health organization (WHO) scale:

  1. Not hospitalized and no COVID-19 related symptoms;
  2. Not hospitalized, with COVID-19 related symptoms;
  3. Hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infection-control or other nonmedical reasons);
  4. Hospitalized, not requiring supplemental oxygen but requiring ongoing medical care (related to COVID-19);
  5. Hospitalized, requiring any supplemental oxygen by nasal cannula;
  6. Hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices;
  7. Hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); and
  8. Death.

     Immunocompromised patient with hematological malignances is defined as:
* Recipients of an allogeneic stem cell transplantation or other form of cell therapy, for example CAR T-cell therapy
* Patients with hematological malignancies who have been in MRD-negative CR for less than 3 years from the completion of their last treatment.
* Patients with hematological malignancies who have been in MRD-negative CR for more than 3 years from the completion of their last therapy and have a peripheral blood CD4 count <200x109cells/liter
* Patients with hematological malignances who are not in MRD-negative CR and are not expected to require anticancer treatment for at least 28 days after the CTLs infusion.

English and non-English speaking patients. Written informed consent and/or signed assent from patient, parent or guardian. Negative pregnancy test in female patients of childbearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of child bearing potential must be willing to use an effective contraceptive measure while on study.

Willingness to comply with the study protocol requirements.

Exclusion criteria:

* Patients receiving systemic steroids at time of enrollment (physiological substitutive therapy s allowed), or who have received ATG --within 14 days or have received donor lymphocyte infusion (DLI) or Campath within 28 days of enrollment.
* Patients with other infections other than COVID-19
* Active acute or chronic GVHD.
* Patients receiving immunosuppressive therapy
* Patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Assessment of feasibility | Up to 3 months post-infusion
  Proportion of patients who receive at least one severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) specific cytotoxic T lymphocytes (CTLs) infusion. Study approach will be considered feasible if at least 50% of the enrolled eligible patients receive one CTLs infusion.
Incidence of adverse events | Up to 3 months post-infusion
  Will collect adverse events and grade them according to Common Terminology Criteria for Adverse Events version 4.0. Attribution will be assigned based on the relationship to the cell infusion.

SECONDARY OUTCOMES:
Response to cytotoxic T lymphocytes | Up to 2 weeks post-infusion
  Defined as extubation for patients who required intubation and mechanical ventilation, reduction in the need of oxygen of 50% or a reduction in the fraction of inspired oxygen (FiO2) below 30% or oxygen discontinuation for patients who are not intubated but require oxygen, or resolution of clinical and radiological signs and symptoms for patients who do not require oxygen. Proportion of patients experiencing response will be computed with associated 95% confidence interval.
Overall survival | From treatment start date to date of death, assessed up to 3 months post-infusion
  Will be estimated using the Kaplan-Meier method.
Relapse free survival (original malignancy) | From treatment start date to the date of documented disease recurrence or death, assessed up to 3 months post-infusion
  Will be estimated using the Kaplan-Meier method.
Cumulative incidence of coronavirus disease 2019 pneumonia resolution after therapy | Up to 3 months post-infusion
Cumulative incidence of grade 2-4 or 3-4 graft versus host disease (GVHD), and chronic GVHD | Up to 3 months post-infusion
  Will be assessed using the competing risks method. The competing risks will include relapse and death and patients who are still alive without disease progression at end of study will be censored.
All-cause mortality | At 28 days post-infusion
Proportion of subjects alive and free of respiratory failure | At 28 days post-infusion
Reconstitution of anti-virus immunity | Up to 3 months post-infusion
  Number of SARS-COV-2 specific T-cells in blood will be determined for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: David Marin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT04742595/ICF_000.pdf